CLINICAL TRIAL: NCT03698292
Title: The Study of The Efficacy and Safety of Itopride For Feeding Intolerance in Critically-ill Patients Receiving Enteral Nutrition
Brief Title: Itopride in Feeding Intolerance of Critically-ill Patients Receiving Enteral Nutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Mohamed El Mokadem, Assistant Lecturer, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 67
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Critically-ill Patients
MeSH Terms: interventions — itopride; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First group (Active Comparator): Metoclopramide 10 mg tablets will be taken by the patients of this group three times daily for 7 days
  Interventions: Drug: Metoclopramide 10mg
- Second Group (Active Comparator): Itopride 50 mg tablets will be taken by the patients of this group three times daily for 7 days
  Interventions: Drug: Itopride

INTERVENTIONS:
Drug: Itopride — Prokinetic Drug
  Arms: Second Group
Drug: Metoclopramide 10mg — Prokinetic Drug
  Arms: First group

SUMMARY:
The current study will compare the effectiveness as well as the safety of Itopride against metoclopramide as the first line treatment for feeding intolerance in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging between 18 and 60 years (of both sexes) who are admitted to the ICU and are expected to stay in the ICU for not less than 7 days and are prescribed enteral feeding through naso- or oro-gastric tube whose modified nutritional risk in the critically ill (mNUTRIC) score is of more than or equal 5.

Exclusion Criteria:

* Patients who met the following criteria were excluded:

  * Age less than 18 years or more than 60 years.
  * Previous upper gastrointestinal tract surgery, obstruction, hemorrhage or history of GI disease.
  * Clinically significant hepatic dysfunction. (>3 times above the upper end of normal range of bilirubin, γ-glutamyl transferase, aspartate transaminase, or lactate dehydrogenase)
  * Regular use of H2 blockers, prokinetic, proton pump inhibitor or anticholinergic agents for previous 4 weeks.
  * Patients with arrhythmia or atrioventricular blocks.
  * Any condition or comorbid disease that might interfere with gastric emptying such as diabetes.
  * Patients with head injuries.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Gastric Residual Volume | 7 days
  Gastric residual volume as a surrogate to gastric emptying by means of gastric ultrasound.
  of the study, at midpoint of the study and at the end of the study by guided ultrasonography.

SECONDARY OUTCOMES:
Determining the adequacy of enteral nutrition | 24 hours
  By calculating the ratio between administered and prescribed feeds over 24 hours duration (Percentage of feed goal tolerated)
Length of ICU stay | 3 months
  Length of patients stay in the ICU will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gholipour Baradari A, Alipour A, Firouzian A, Moarab L, Emami Zeydi A. A Double-Blind Randomized Clinical Trial Comparing the Effect of Neostigmine and Metoclopramide on Gastric Residual Volume of Mechanically Ventilated ICU Patients. Acta Inform Med. 2016 Dec;24(6):385-389. doi: 10.5455/aim.2016.24.385-389. PMID 28077899
- [Background] Gomes PC, Caporossi C, Aguilar-Nascimento JE, Silva AM, Araujo VM. Residual gastric volume evaluation with ultrasonography after ingestion of carbohydrate- or carbohydrate plus glutamine-enriched beverages: a randomized, crossover clinical trial with healthy volunteers. Arq Gastroenterol. 2017 Jan-Mar;54(1):33-36. doi: 10.1590/S0004-2803.2017v54n1-06. PMID 28079236
- [Derived] Elmokadem EM, El Borolossy RM, Bassiouny AM, Hanna MG, Darweesh EAG, Sabri NA. The efficacy and safety of itopride in feeding intolerance of critically ill patients receiving enteral nutrition: a randomized, double-blind study. BMC Gastroenterol. 2021 Mar 19;21(1):126. doi: 10.1186/s12876-021-01712-w. PMID 33740892